CLINICAL TRIAL: NCT06794801
Title: An Open-Label, Prospective, Single-Center, Randomized Controlled Trial Evaluating the Safety and Efficacy of Drug-Coated Autoperfusion Balloons Versus Conventional Drug-Coated Balloons Guided by IVUS-OCT Multimodal Imaging for Treating Acute Myocardial Infarction: OPERA-AMI Study
Brief Title: Evaluating the Safety and Efficacy of Drug-Coated Autoperfusion Balloons Versus Conventional Drug-Coated Balloons Guided by IVUS-OCT Multimodal Imaging for Treating Acute Myocardial Infarction: OPERA-AMI Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LanZhou University (Other)
Responsible Party: Principal Investigator, BAI MING, MD, LanZhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LLYY2024PJ171
Record Dates: First submitted 2025-01-16; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: ST Segment Elevation Myocardial Infarction (STEMI)
Keywords: Drug Coated Autoperfusion Balloon Dilatation Catheter; Percutaneous Coronary Intervention; VUS-OCT Multimodal Imaging; De novo lesion
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Masking Description: Using a core laboratory, an impartial third-party evaluation will be carried out for this study to objectively assess each participant's intravascular imaging and coronary angiography results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug Coated Autoperfusion Balloon Dilatation Catheter（DCAB） (Experimental): 3 μg/mm² paclitaxel-coated drug-coated autoperfusion balloon dilatation catheter (DCAB). The DCAB features two radiopaque marker rings at the balloon shoulders for intravascular imaging and positioning, self-perfusion holes on the catheter shaft, and an additional radiopaque marker ring proximal to the perfusion holes to indicate their location. The catheter shaft is hydrophilically coated to facilitate blood flow through the perfusion holes when the guidewire is retracted. Preclinical studies show this design allows 15%-20% of arterial blood to reach the distal coronary artery.
  Interventions: Device: Drug Coated Autoperfusion Balloon Dilatation Catheter（DCAB）
- Conventional Drug coated ballon（DCB） (Active Comparator): Bingo® PTCA Drug Delivery System: drug (paclitaxel) coated balloon (DCB) with concentration of 3 μg Paclitaxel per 1 mm2.
  Interventions: Device: Conventional Drug coated balloon (DCB)

INTERVENTIONS:
Device: Drug Coated Autoperfusion Balloon Dilatation Catheter（DCAB） — In the experimental arm, under the assessment and guidance of IVUS-OCT, STEMI patients with successfully prepared lesions will be treated with a drug-coated autoperfusion balloon dilatation catheter (DCAB). Successful lesion preparation is defined as post-pretreatment residual stenosis ≤ 30%, no type C dissections, intravascular imaging confirming no significant residual plaque burden at the dissection site, no transverse expansion > 60°, no longitudinal expansion > 2 mm, no dissection involving the media or adventitia, and no location at the stent distal end. There should be no hematoma and no significant thrombus (TIMI thrombus burden grade ≤ 2). If the angiographic and intravascular imaging results after DCAB treatment are unsatisfactory, an emergency drug-eluting stent (DES) will be implanted.
  Arms: Drug Coated Autoperfusion Balloon Dilatation Catheter（DCAB）
Device: Conventional Drug coated balloon (DCB) — In the control arm, under the assessment and guidance of IVUS-OCT, STEMI patients with successful lesion preparation (residual stenosis ≤ 30%, no type C dissections, no significant residual plaque burden, no dissection involving the media or adventitia, no transverse expansion > 60°, no longitudinal expansion > 2 mm, no location at the stent distal end, no hematoma, TIMI thrombus burden grade ≤ 2) will be treated with a conventional DCB coated with 3 μg/mm2 paclitaxel. If angiographic and intravascular imaging results are unsatisfactory, a bailout DES will be implanted.
  Other Names: Bingo® PTCA Drug Delivery System
  Arms: Conventional Drug coated ballon（DCB）

SUMMARY:
Trial Goals:

1. Evaluation of Mid- to Long-Term Safety and Effectiveness of Drug-Coated Autoperfusion Balloon Dilatation Catheter (DCAB) versus Conventional Drug coated balloon (DCB) in Patients with ST Segment Elevation Myocardial Infarction (STEMI).
2. Evaluation of Hybrid IVUS-OCT System for Intraoperative Evaluation of DCAB or Conventional DCB Treatment Safety and Effectiveness for De Novo Lesions During Emergency Percutaneous Coronary Intervention (PCI) in Patients with STEMI.

The primary outcome is late lumen loss (LLL) assessed at 9 months following emergency PCI, measured using quantitative coronary angiography (QCA).

ELIGIBILITY:
Inclusion Criteria:

1. Acute ST-Elevation Myocardial Infarction Meeting PPCI Criteria: 1) Chest pain lasting more than 20 minutes, with ST-segment elevation of at least 1 mm in two or more adjacent leads, new left bundle branch block, or evidence of posterior wall myocardial infarction; 2) Onset of symptoms within 12 hours.
2. Patients Who Have Received Thrombolytic Therapy Within 6 Hours of Symptom Onset and Are Eligible for Rescue PCI Within 24 Hours;
3. Infarct-Related Artery Selection Imaging and Pre-Treatment Criteria Meeting PPCI Standards: 1) De novo lesions. 2) Reference vessel diameter between 2.5 mm and 4 mm. 3) Successful pre-treatment of target lesions: post-pre-treatment residual stenosis of the culprit vessel ≤ 30%, with no type C dissections (or intravascular imaging indicating significant residual plaque burden at the site of dissection, with transverse expansion > 60°, longitudinal expansion > 2 mm, dissection involving the media or adventitia, and located at the distal end of the stent), no hematoma, and no significant thrombus (TIMI thrombus burden grade ≤ 2);
4. Sufficient compliance with the study protocol, agreement to undertake follow-up, and coronary angiography at 9 months;
5. Voluntary Participation in This Study, Including Signing a Written Informed Consent with Understanding of All Risks and Benefits Described in the Informed Consent Document.

Exclusion Criteria:

1. Age < 18 years and > 75 years;
2. History of prior myocardial infarction;
3. Allergy to contrast agent/inability to tolerate contrast;
4. Known contraindications / inability to tolerate bivalirudin, fondaparinux, heparin, aspirin, clopidogrel, and/or ticagrelor;
5. Complex coronary lesions: left main lesions, lesions at the ostia of the left anterior descending or circumflex arteries, lesion length > 30 mm, severe calcification, severe tortuosity or angulation, bifurcation lesions requiring the implantation of more than two drug-coated balloons (DCBs) or drug-eluting stents;
6. In-stent restenosis or in-stent thrombus lesions;
7. Planned simultaneous intervention on non-target lesions;
8. Active bleeding or recent history of bleeding;
9. Uncertain neurological outcomes, such as resuscitation;
10. Intubation / ventilation;
11. Cardiogenic shock prior to randomization;
12. Known intracranial disease (tumors, aneurysms, arteriovenous malformations, hemorrhagic CVA, ischemic CVA/TIA within the last 6 months, including permanent neurological deficits from ischemic cerebrovascular disease) ;
13. Refusal of blood transfusion;
14. Planned major surgery within 6 weeks;
15. Stent implantation < 1 month prior to enrollment;
16. Life expectancy of less than 12 months;
17. Participation in another clinical trial that interferes with this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Late lumen loss at 9 months after index PCI | 9±2 months
  Late lumen loss, as assessed by quantitative coronary angiography, at 9 months following the index percutaneous coronary intervention.

SECONDARY OUTCOMES:
Incidence of patient-oriented composite endpoint (PoCE) | 3±1 Months, 6±1 Months, 9±2 Months, 2 Years, 3 Years, 4 Years, and 5 Years after PCI
  Incidence of patient-oriented composite endpoint (PoCE) and individual components of PoCE: defined as a composite of all-cause death, Target vessel failure, any stroke, any myocardial infarction (MI), and any clinically or physiologically indicated revascularization.
Incidence of Bleeding Academic Research Consortium bleeding type 3 and 5 bleeding complications | 3±1 Months, 6±1 Months, 9±2 Months, 2 Years, 3 Years, 4 Years, and 5 Years after PCI
  Bleeding Academic Research Consortium type 3 and 5 bleeding complications
Incidence of coronary dissection, categorized by Types A, B, C, and D-F, immediately following DCB implantation | index PCI
  Based on the results of coronary angiography after DCB implantation
The incidence of bailout stenting following DCB implantation | index PCI
  The following criteria are used to define it: TIMI flow ≤ Grade 2; residual stenosis > 30%; Type C (or intravascular imaging demonstrating significant residual plaque burden at the dissection site, lateral extension > 60°, longitudinal extension > 2 mm, dissection involving the media or adventitia); and higher dissection.
Minimum lumen area and Lumen Area Loss Immediately After DCB Implantation by IVUS-OCT Intravascular Imaging. | index PCI
  Change in minimum lumen area and lumen area loss (in mm2), as assessed by IVUS-OCT multimodal imaging, compared with pre-procedure baseline following coronary artery drug-coated balloon angioplasty.
Incidence of intolerable adverse events during the duration of coronary artery drug-coated balloon dilation. | index PCI
  Incidence of intolerable worsening chest pain, hemodynamic instability, ST-segment changes, and severe arrhythmias during DCB expansion and duration of DCB expansion.

CONTACTS AND LOCATIONS:
Locations (1):
- LanZhou University, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: Yes
The data is available and can be requested, subject to approval, if a reasonable clinical research analysis plan is provided to the corresponding author.
Supporting Information: CSR
Time Frame: 6 months
Access Criteria: Submit a detailed research analysis plan to the corresponding author and apply through our email.
URL: https://www.lzdxdyyy.com/Web/Ldyy

REFERENCES:
- [Background] Keeley EC, Boura JA, Grines CL. Primary angioplasty versus intravenous thrombolytic therapy for acute myocardial infarction: a quantitative review of 23 randomised trials. Lancet. 2003 Jan 4;361(9351):13-20. doi: 10.1016/S0140-6736(03)12113-7. PMID 12517460
- [Background] Grines CL, Cox DA, Stone GW, Garcia E, Mattos LA, Giambartolomei A, Brodie BR, Madonna O, Eijgelshoven M, Lansky AJ, O'Neill WW, Morice MC. Coronary angioplasty with or without stent implantation for acute myocardial infarction. Stent Primary Angioplasty in Myocardial Infarction Study Group. N Engl J Med. 1999 Dec 23;341(26):1949-56. doi: 10.1056/NEJM199912233412601. PMID 10607811
- [Background] Suryapranata H, van 't Hof AW, Hoorntje JC, de Boer MJ, Zijlstra F. Randomized comparison of coronary stenting with balloon angioplasty in selected patients with acute myocardial infarction. Circulation. 1998 Jun 30;97(25):2502-5. doi: 10.1161/01.cir.97.25.2502. PMID 9657469
- [Background] Serruys PW, Degertekin M, Tanabe K, Abizaid A, Sousa JE, Colombo A, Guagliumi G, Wijns W, Lindeboom WK, Ligthart J, de Feyter PJ, Morice MC; RAVEL Study Group. Intravascular ultrasound findings in the multicenter, randomized, double-blind RAVEL (RAndomized study with the sirolimus-eluting VElocity balloon-expandable stent in the treatment of patients with de novo native coronary artery Lesions) trial. Circulation. 2002 Aug 13;106(7):798-803. doi: 10.1161/01.cir.0000025585.63486.59. PMID 12176950
- [Background] McFadden EP, Stabile E, Regar E, Cheneau E, Ong AT, Kinnaird T, Suddath WO, Weissman NJ, Torguson R, Kent KM, Pichard AD, Satler LF, Waksman R, Serruys PW. Late thrombosis in drug-eluting coronary stents after discontinuation of antiplatelet therapy. Lancet. 2004 Oct 23-29;364(9444):1519-21. doi: 10.1016/S0140-6736(04)17275-9. PMID 15500897
- [Background] Brott BC, Anayiotos AS, Chapman GD, Anderson PG, Hillegass WB. Severe, diffuse coronary artery spasm after drug-eluting stent placement. J Invasive Cardiol. 2006 Dec;18(12):584-92. PMID 17197707
- [Background] Nakazawa G, Finn AV, Joner M, Ladich E, Kutys R, Mont EK, Gold HK, Burke AP, Kolodgie FD, Virmani R. Delayed arterial healing and increased late stent thrombosis at culprit sites after drug-eluting stent placement for acute myocardial infarction patients: an autopsy study. Circulation. 2008 Sep 9;118(11):1138-45. doi: 10.1161/CIRCULATIONAHA.107.762047. Epub 2008 Aug 25. PMID 18725485
- [Background] Vink MA, Dirksen MT, Suttorp MJ, Tijssen JG, van Etten J, Patterson MS, Slagboom T, Kiemeneij F, Laarman GJ. 5-year follow-up after primary percutaneous coronary intervention with a paclitaxel-eluting stent versus a bare-metal stent in acute ST-segment elevation myocardial infarction: a follow-up study of the PASSION (Paclitaxel-Eluting Versus Conventional Stent in Myocardial Infarction with ST-Segment Elevation) trial. JACC Cardiovasc Interv. 2011 Jan;4(1):24-9. doi: 10.1016/j.jcin.2010.11.003. PMID 21251625
- [Background] Gonzalo N, Barlis P, Serruys PW, Garcia-Garcia HM, Onuma Y, Ligthart J, Regar E. Incomplete stent apposition and delayed tissue coverage are more frequent in drug-eluting stents implanted during primary percutaneous coronary intervention for ST-segment elevation myocardial infarction than in drug-eluting stents implanted for stable/unstable angina: insights from optical coherence tomography. JACC Cardiovasc Interv. 2009 May;2(5):445-52. doi: 10.1016/j.jcin.2009.01.012. PMID 19463469
- [Background] Ali RM, Abdul Kader MASK, Wan Ahmad WA, Ong TK, Liew HB, Omar AF, Mahmood Zuhdi AS, Nuruddin AA, Schnorr B, Scheller B. Treatment of Coronary Drug-Eluting Stent Restenosis by a Sirolimus- or Paclitaxel-Coated Balloon. JACC Cardiovasc Interv. 2019 Mar 25;12(6):558-566. doi: 10.1016/j.jcin.2018.11.040. PMID 30898253
- [Background] Jeger RV, Farah A, Ohlow MA, Mangner N, Mobius-Winkler S, Weilenmann D, Wohrle J, Stachel G, Markovic S, Leibundgut G, Rickenbacher P, Osswald S, Cattaneo M, Gilgen N, Kaiser C, Scheller B; BASKET-SMALL 2 Investigators. Long-term efficacy and safety of drug-coated balloons versus drug-eluting stents for small coronary artery disease (BASKET-SMALL 2): 3-year follow-up of a randomised, non-inferiority trial. Lancet. 2020 Nov 7;396(10261):1504-1510. doi: 10.1016/S0140-6736(20)32173-5. Epub 2020 Oct 19. PMID 33091360
- [Background] Jeger RV, Eccleshall S, Wan Ahmad WA, Ge J, Poerner TC, Shin ES, Alfonso F, Latib A, Ong PJ, Rissanen TT, Saucedo J, Scheller B, Kleber FX; International DCB Consensus Group. Drug-Coated Balloons for Coronary Artery Disease: Third Report of the International DCB Consensus Group. JACC Cardiovasc Interv. 2020 Jun 22;13(12):1391-1402. doi: 10.1016/j.jcin.2020.02.043. Epub 2020 May 27. PMID 32473887
- [Background] Vos NS, Dirksen MT, Vink MA, van Nooijen FC, Amoroso G, Herrman JP, Kiemeneij F, Patterson MS, Slagboom T, van der Schaaf RJ. Safety and feasibility of a PAclitaxel-eluting balloon angioplasty in Primary Percutaneous coronary intervention in Amsterdam (PAPPA): one-year clinical outcome of a pilot study. EuroIntervention. 2014 Sep;10(5):584-90. doi: 10.4244/EIJV10I5A101. PMID 25256200
- [Background] Laarman GJ, Suttorp MJ, Dirksen MT, van Heerebeek L, Kiemeneij F, Slagboom T, van der Wieken LR, Tijssen JG, Rensing BJ, Patterson M. Paclitaxel-eluting versus uncoated stents in primary percutaneous coronary intervention. N Engl J Med. 2006 Sep 14;355(11):1105-13. doi: 10.1056/NEJMoa062598. PMID 16971717
- [Background] Kastrati A, Dibra A, Spaulding C, Laarman GJ, Menichelli M, Valgimigli M, Di Lorenzo E, Kaiser C, Tierala I, Mehilli J, Seyfarth M, Varenne O, Dirksen MT, Percoco G, Varricchio A, Pittl U, Syvanne M, Suttorp MJ, Violini R, Schomig A. Meta-analysis of randomized trials on drug-eluting stents vs. bare-metal stents in patients with acute myocardial infarction. Eur Heart J. 2007 Nov;28(22):2706-13. doi: 10.1093/eurheartj/ehm402. Epub 2007 Sep 27. PMID 17901079
- [Background] Kim HS, Lee JH, Lee SW, Kim YH, Park JH, Choi SW, Jeong JO, Seong IW, Rhee KS, Ko JK, Jo SH, Choi YJ. Long-term safety and efficacy of sirolimus- vs. paclitaxel-eluting stent implantation for acute ST-elevation myocardial infarction: 3-year follow-up of the PROSIT trial. Int J Cardiol. 2011 Mar 3;147(2):253-7. doi: 10.1016/j.ijcard.2009.09.466. Epub 2009 Sep 26. PMID 19783056
- [Background] Vos NS, Fagel ND, Amoroso G, Herrman JR, Patterson MS, Piers LH, van der Schaaf RJ, Slagboom T, Vink MA. Paclitaxel-Coated Balloon Angioplasty Versus Drug-Eluting Stent in Acute Myocardial Infarction: The REVELATION Randomized Trial. JACC Cardiovasc Interv. 2019 Sep 9;12(17):1691-1699. doi: 10.1016/j.jcin.2019.04.016. Epub 2019 May 21. PMID 31126887
- [Background] Gao C, He X, Ouyang F, Zhang Z, Shen G, Wu M, Yang P, Ma L, Yang F, Ji Z, Wang H, Wu Y, Fang Z, Jiang H, Wen S, Liu Y, Li F, Zhou J, Zhu B, Liu Y, Zhang R, Zhang T, Wang P, Liu J, Jiang Z, Xia J, van Geuns RJ, Capodanno D, Garg S, Onuma Y, Wang D, Serruys PW, Tao L; REC-CAGEFREE I Investigators. Drug-coated balloon angioplasty with rescue stenting versus intended stenting for the treatment of patients with de novo coronary artery lesions (REC-CAGEFREE I): an open-label, randomised, non-inferiority trial. Lancet. 2024 Sep 14;404(10457):1040-1050. doi: 10.1016/S0140-6736(24)01594-0. Epub 2024 Sep 2. PMID 39236727
- [Background] Hao X, Huang D, Wang Z, Zhang J, Liu H, Lu Y. Correction to: Study on the safety and effectiveness of drug-coated balloons in patients with acute myocardial infarction. J Cardiothorac Surg. 2021 Sep 3;16(1):247. doi: 10.1186/s13019-021-01629-1. No abstract available. PMID 34474673